CLINICAL TRIAL: NCT01263860
Title: A Randomized Trial of 24-Week Versus 48-Week Courses of Peginterferon Plus
Brief Title: A Randomized Trial of 24-Week Versus 48-Week Courses of Peginterferon Plus Ribavirin for HCV Genotype-6 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cai Qingxian, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAH115G6HCV
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24-Week treatment group (Experimental): Genotype 6 chronic hepatitis C patients with rapid virological response(undetectable HCV RNA at weeks 4) in this group will be treated with Peginterferon alfa-2a plus ribavirin for an additional 20 weeks
  Interventions: Drug: Peginterferon alfa2a; Drug: Ribavirin
- 48-Week treatment group (Active Comparator): Genotype 6 chronic hepatitis C patients with rapid virological response(undetectable HCV RNA at weeks 4) in this group will be treated with Peginterferon alfa-2a plus ribavirin for an additional 44 weeks
  Interventions: Drug: Peginterferon alfa2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa2a — patients receive a dose of 180 µg of PEGASYS once a week for 24 weeks
  Arms: 24-Week treatment group
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 24 weeks
  Arms: 24-Week treatment group
Drug: Peginterferon alfa2a — patients receive a dose of 180 µg of PEGASYS once a week for 48 weeks
  Arms: 48-Week treatment group
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 48 weeks
  Arms: 48-Week treatment group

SUMMARY:
Patients with HCV genotype 6 infection who have a rapid virological response to treatment are randomised to either 24 or 48 weeks HCV treatment. Our hypothesis is that there is no important difference in effect between the two treatment effect.

DETAILED DESCRIPTION:
High rate of infection of Hepatitis C Virus(HCV) Genotype 6 was recently confirmed in Southern China. Recent study implied chronic hepatitis C genotype 6 responds better to the 48-week treatment with pegylated interferon and ribavirin than genotype 1. Approximately 75.7% obtain sustained virological response (HCV RNA undetectable 24 weeks after treatment) to this approach. However, the treatment is associated with many and sometimes serious side effects. In addition, the treatment is costly also in economical terms. Shorter treatment for chronic hepatitis C genotype 6 is necessary to be assessed.

In this randomised,open label,multicenter phase 3 trial with active controls patients are treated with pegylated interferon alfa 2a (180ug/week)and ribavirin(800-1200mg based on weight)for 4 weeks. Those who are HCV RNA negative at week 4 (<50 IU; Cobas Amplicor Monitor Test, Roche Diagnostic) are defined as rapid virological responders and randomised to either an additional 20 or 44 weeks combination treatment. Patients who are HCV RNA positive are all treated for 44 more weeks. The endpoint is sustained virological response defined as undetectable HCV RNA 24 weeks after end of treatment.

Our hypothesis is that there is no important difference in the effect in the two groups.

This is a non-inferiority trial. The smallest difference considered to be clinically important is 15%. Thus to state "non-inferiority" the 95% confidence interval of the observed difference between the groups shall not overlap 10%. Both intention to treat and and per protocol analyses will be published. Conclusion will be conservative and based on the analysis who detect the biggest difference.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA is positive
* Genotype 6
* Treatment naive
* Raised ALT

Exclusion Criteria:

* Active substance abuse
* Poorly controlled psychiatric disease
* HBsAg positive
* Anti-HIV positive
* Suffering from other significant concurrent medical conditions including chronic liver diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 weeks after the end of treatment
  Undetectable HCVRNA in serum(<15IU/ml) 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Change in health related quality as measured by short from 36 (SF-36) from baseline to 24 weeks after the end of treatment | 24 weeks after the end of treatment
Sick leave in patients treated for 24 or 48 weeks treatment | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gao Zhiliang, Doctor, Study Chair — The Third Affliated Hospital of Sun Yat-sen University; Zhao Zhixin, Doctor, Study Director — The Third Affliated Hospital of Sun Yat-sen University; Zhang Xiaohong, Doctor, Principal Investigator — The Third Affliated Hospital of Sun Yat-sen University; Xu Min, Doctor, Principal Investigator — The Eighth People's Hospital of Guangzhou; Wei min, Doctor, Principal Investigator — Zhongshan second people's hospital; Huang mingshou, Bachelor, Principal Investigator — Panyu People's Hospital
Locations (4):
- China (4):
  - The Eighth People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Panyu People's Hospital, Guangzhou, Guangdong
  - Zhongshan second people's hospital, Zhongshan, Guangdong

REFERENCES:
- [Derived] Cai Q, Zhang X, Lin C, Shao X, Guan Y, Deng H, Wei M, Huang M, Ren Z, Lu L, Mei Y, Xu M, Zhu J, Shi H, Lin G, Liu Y, Hu F, Luo Q, Lan Y, Guo F, Zhao Z, Gao Z. 24 versus 48 Weeks of Peginterferon Plus Ribavirin in Hepatitis C Virus Genotype 6 Chronically Infected Patients with a Rapid Virological Response: A Non-Inferiority Randomized Controlled Trial. PLoS One. 2015 Oct 28;10(10):e0140853. doi: 10.1371/journal.pone.0140853. eCollection 2015. PMID 26509605